CLINICAL TRIAL: NCT00075621
Title: A Phase II Trial of Tandem Transplantation in AL Amyloidosis
Brief Title: Tandem Autologous Stem Cell Transplantation in Treating Patients With Primary Systemic (AL) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23645
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- tandem transplant (Other): Drug: filgrastim 16 mg/kg/day for 3 days prior to stem cell collection, through day before last collection
  Drug: melphalan 200 mg/kg over 2 days
  Procedure/Surgery: autologous peripheral blood stem cell transplantation
  autologous peripheral blood stem cell transplantation
  Interventions: Drug: filgrastim; Drug: melphalan; Procedure: autologous peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: filgrastim — 16 mg/kg/day for 3 days prior to stem cell collection, through day before last collection
Drug: melphalan — 200 mg/kg over 2 days
  Other Names: alkeran
Procedure: autologous peripheral blood stem cell transplantation — autologous peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Autologous stem cell transplantation may be effective treatment for primary systemic (AL) amyloidosis.

PURPOSE: This phase II trial is studying how well tandem (two) autologous stem cell transplantation works in treating patients with primary systemic (AL) amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerability of tandem autologous stem cell transplantation in patients with AL amyloidosis.
* Determine whether this regimen can convert a hematologic non-complete response (CR) to CR in these patients.
* Determine the overall survival of patients treated with this regimen.

OUTLINE:

* First transplantation: Patients receive filgrastim (G-CSF) subcutaneously once daily beginning 3 days before the initiation of stem cell collection and continuing until the day before the completion of stem cell collection. Patients may undergo bone marrow harvest if an inadequate number of peripheral blood stem cells are collected.

Patients receive high-dose melphalan IV over 20 minutes on days -3 and -2. Patients undergo autologous stem cell transplantation (ASCT) on day 0.

* Second transplantation: Within 6-12 months after the first ASCT, patients not achieving a complete response receive high-dose melphalan IV over 20 minutes on days -3 and -2 and a second ASCT on day 0.

Treatment continues in the absence of unacceptable toxicity.

Patients are followed at 3 and 6 months, 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed AL amyloidosis, meeting 1 of the following criteria:

  * Plasma cell dyscrasia, evidenced by 1 of the following:

    * Monoclonal protein in the serum or urine by immunofixation electrophoresis
    * Plasmacytosis of the bone marrow with monoclonal staining for kappa or lambda light chain isotype
  * Macroglossia with at least 1 other site having biopsy proven amyloidosis and absence of a mutant transthyretin is ruled out

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* SWOG 0-2

Life expectancy

* At least 1 year

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* LVEF ≥ 45% by MUGA or echocardiogram

Pulmonary

* DLCO ≥ 50%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to tolerate 2 courses of high-dose therapy
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior alkylating agent chemotherapy allowed provided there is no morphologic or cytogenetic evidence of myelodysplastic syndromes
* Prior total cumulative oral melphalan dose < 300 mg

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior cytotoxic therapy and recovered

Exclusion Criteria:

* No senile, secondary, localized, dialysis-related, or familial amyloidosis
* No overt multiple myeloma (e.g., greater than 30% bone marrow plasmacytosis, extensive [more than 2] lytic lesions, hypercalcemia)

Cardiovascular

* No myocardial infarction within the past 6 months
* No congestive heart failure
* No arrhythmia refractory to therapy
* No evidence of symptomatic transient ischemic attacks or strokes
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2000-08 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
safety | 100 days, 6 months, and annual

SECONDARY OUTCOMES:
Efficacy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Cancer Research Center at Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No